CLINICAL TRIAL: NCT06100510
Title: PFA 100 Evaluation and Reference Interval HOACNY
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Hematology Oncology Associates of Central New York (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HOACNYPFA100.001
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (non-intervention) Arm (No Intervention): Participants who will have PFA 100 testing performed without the ingestion of aspirin.
- Aspirin Arm (Active Comparator): Participants who will have PFA 100 testing performed after the ingestion of aspirin.
  Interventions: Drug: Aspirin 325mg

INTERVENTIONS:
Drug: Aspirin 325mg — Cohort B will receive one (1) 325 mg aspirin 24 hours prior to their second blood draw.
  Arms: Aspirin Arm

SUMMARY:
The purpose of this research is to evaluate instrument functionality and develop a reference range of normal data by healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to consent to study

Exclusion Criteria from entire study

* Primary hemostasis diagnosis

  * Von Willebrand Disease
  * Bernard-Soulier syndrome
  * Glanzmann thrombasthenia
  * Idiopathic thrombocytopenic purpura
  * Drug-induced thrombocytopenia
  * Heparin-induced thrombocytopenia
  * Thrombotic thrombocytopenic purpura
  * Hemolytic uremic syndrome
* Participant is on anticoagulant therapy

  * Specifically thienopyrdines [Ticlopidine, Clopidogrel] and GPIIb/IIIa inhibitors [ReoPro, Aggrastat, Integrilin]
* Participant is on medication that contains ASA or aspirin (see list below in Study Procedure)
* Participant is on nonsteroidal anti-inflammatory agents that are known to induce temporary platelet dysfunction (see list below in Study Procedure)
* Participant is on non-prescription medications containing aspirin (see list below in Study Procedure)
* PFA-100 result falls outside of reference interval listed in the package insert (suggested criteria in the PFA-100 Evaluation Protocol as described in the PFA-100 System: Getting Started Guide)
* If hematocrit is less than 35%
* If platelets are less than 150 x10^3/uL

Exclusion Criteria from Cohort B but not Cohort A

* Potential for adverse reactions between current medication and aspirin as dictated by staff pharmacist
* Allergy to ASA or aspirin
* Previous allergic reaction to ASA or aspirin
* Participant is pregnant
* Asthma, or history of, with nasal polyps and rhinitis
* Stomach ulcers or bleeding
* Severe kidney disease
* Severe liver disease
* Hemophilia
* Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Instrument Evaluation Protocol-PFA100 Instrumentation [platelet function as measured by aperture closure time monitored in seconds for collagen/epinephrine (COL/EPI) cartridges and collagen/ADP (COL/ADP) cartridges] | 3 months
  This portion of the study is to ensure that the functionality of the instrumentation is working properly.
  For each participant, their pre-aspirin dose closure times will be compared to their post-aspirin dose closure times.
  The typical pattern seen in subjects with normal platelet function (pre-aspirin testing) is closure time (CT) results within the reference range for both the COL/EPI and COL/ADP cartridges (normal).
  In general, the pattern seen after aspirin ingestion is a CT result outside the reference range (abnormal) with COL/EPI and within the reference range for COL/ADP (normal).
Reference Interval Protocol-PFA100 Instrumentation [platelet function as measured by aperture closure time monitored in seconds for collagen/epinephrine (COL/EPI) cartridges and collagen/ADP (COL/ADP) cartridges] | 3 months
  For each participant in the non-intervention/placebo arm, platelet function as measured by aperture closure time monitored in seconds for collagen/epinephrine (COL/EPI) cartridges and collagen/ADP (COL/ADP) cartridges will be captured.
  Following guidelines as stated per CLSI document EP28-A3c, a reference interval will be developed from this captured data.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa O'Sullivan, BS,MLT(ASCP), Principal Investigator — Employee; Steven Duffy, MD, Study Director — Physician
Locations (1):
- Hematology Oncology Associates of Central New York, East Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.